CLINICAL TRIAL: NCT05187377
Title: Electrophysiological Markers for Interventions in Phelan-McDermid Syndrome and Idiopathic Autism
Brief Title: A Controlled Trial of Growth Hormone in Phelan-McDermid Syndrome and Idiopathic Autism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Alexander Kolevzon, Clinical Director, Seaver Autism Center for Research & Treatment, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY-18-00245; R01NS105845 (NIH); GCO 17-1159 (Other: Icahn School of Medicine at Mount Sinai)
Record Dates: First submitted 2021-12-28; First posted 2022-01-11 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Phelan-McDermid Syndrome; Autism Spectrum Disorder (ASD)
Keywords: Autism Spectrum Disorder; Phelan-McDermid Syndrome; 22q13 deletion Syndrome; Growth Hormone; Insulin-Like Growth Factor-1; Electrophysiology
MeSH Terms: conditions — Telomeric 22q13 Monosomy Syndrome; Autism Spectrum Disorder | interventions — Growth Hormone; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled, crossover design, with 12 weeks in each treatment phase (rhGH and placebo) and a four week wash-out period between phases.
  During each phase, participants will be monitored at Baseline, Week 2, Week 4, Week 8, and Week 12.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Mount Sinai Pharmacy will be responsible for randomizing research participants and preparing investigational drug/placebo. The participant, caregivers, and study team will all remain blinded for the duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Growth Hormone then Saline (Experimental): 12 weeks in each treatment phase (rhGH then placebo) and a four week wash-out period between phases.
  Interventions: Drug: Growth Hormone
- Placebo (saline) then Growth Hormone (Placebo Comparator): 12 weeks in each treatment phase (placebo then rhGH) and a four week wash-out period between phases.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Growth Hormone — Growth hormone will be administered subcutaneously once daily. A starting dose of 0.15 mg/kg/week divided daily for 2 weeks to ensure safety and tolerance. The dose will then be increased to 0.3 mg/kg/week for 10 weeks. Doses will be titrated based on IGF-1 levels and monitored every four weeks up to a maximum dose of 0.45 mg/kg/week based on the package insert.
  Other Names: rhGH
  Arms: Growth Hormone then Saline
Drug: Saline — Placebo (saline) will be administered subcutaneously once daily.
  Other Names: placebo
  Arms: Placebo (saline) then Growth Hormone

SUMMARY:
This clinical trial will use growth hormone as a novel treatment for Phelan-McDermid syndrome (PMS) and idiopathic autism. A double-blind, placebo-controlled crossover trial design will be used in 30 children with idiopathic autism and 15 children with PMS to evaluate the the effects of growth hormone on visual evoked potentials (VEPs), socialization, language, and repetitive behaviors. The researchers expect to provide evidence for the feasibility of using VEPs in PMS, and to show support for growth hormone in ameliorating clinical symptoms of ASD.

DETAILED DESCRIPTION:
This study will show that select electrophysiological markers in PMS are relevant to iASD and predictive of treatment response with growth hormone. The long-term goal is to optimize treatment selection in iASD by establishing biological signature(s) derived from PMS. The expected outcome is to establish the feasibility of electrophysiological biomarkers for use in clinical trials in PMS and iASD, demonstrate efficacy of growth hormone in PMS and iASD, and to define a biological profile that will mark a subset of patients with iASD likely to show clinical response to growth hormone.

The study will enroll 45 children (15 PMS; 30 iASD; age 2-12 years) and administer growth hormone/placebo as once daily subcutaneous injection for 12 weeks at standard doses. The study team will monitor baseline anthropometric measures, laboratory parameters for growth, IGF-1 levels, and bone age throughout the study. Evaluations will include validated behavioral scales. Visual evoked potentials (VEPs) will be used as biomarkers of visual sensory reactivity.

Growth Hormone is approved by the FDA for the treatment of children with short stature due to primary growth hormone deficiency, among several other indications. It is being used off-label in the current study and is not FDA approved for use in PMS or ASD.

ELIGIBILITY:
Inclusion Criteria:

* Children between 2 and 12 years of age
* Open epiphyses on bone age x ray
* Must be on stable medication and psychosocial treatment regimens for at least three months prior to enrollment, assuming the concomitant medication is safe for use with Growth Hormone
* No prior use of Growth Hormone or IGF-1
* ASD group: Meet DSM-5 criteria for Autism Spectrum Disorder confirmed by the Autism Diagnostic Interview-Revised (ADI-R) and the Autism Diagnostic Observation Schedule, Second Edition (ADOS-2); absence of known pathogenic copy number variants
* PMS group: Known pathogenic deletions or mutations in SHANK3 gene diagnosed by array CGH and/or direct sequencing

Exclusion Criteria:

* Closed epiphyses
* Active or suspected neoplasia
* Intracranial hypertension
* Hepatic insufficiency
* Renal insufficiency
* Cardiomegaly/valvulopathy
* History of allergy to growth hormone or any component of the formulation (mecasermin)
* Patients with comorbid conditions who are deemed too medically compromised to tolerate the risk of experimental treatment with growth hormone (including severe obesity, sleep apnea, and various acute health conditions)
* Visual problems that preclude the use of VEP

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Visual Evoked Potentials (VEP) | After 12 weeks of growth hormone therapy
  A noninvasive technique to evaluate the functional integrity of visual pathways in the brain from the retina to the visual cortex via the optic nerve/optic radiations. The VEP is recorded from the head's surface, over the visual cortex, and is extracted from ongoing EEG through signal averaging. VEPs reflect the sum of excitatory and inhibitory postsynaptic potentials occurring on apical dendrites which modulate excitatory and inhibitory signals received by the pyramidal cells.

SECONDARY OUTCOMES:
Aberrant Behavior Checklist (ABC) Social Withdrawal Subscale | After 12 weeks of growth hormone therapy
  A caregiver report symptom checklist. 58-item instrument into 5 subscales: Irritability (score 0-45); Lethargy/Social Withdrawal (score 0-48); Stereotypic Behavior (score 0-21); Hyperactivity (score 0-48); Inappropriate Speech (score 0-12). Total scale 0-174, with higher score indicating more aberrant behavior.
Repetitive Behavior Scale-Revised (RBS-R) | After 12 weeks of growth hormone therapy
  A 43 item instrument with total score from 0-129, with higher score indicating more restricted, repetitive and stereotyped behaviors.
Sensory Profile | After 12 weeks of growth hormone therapy
  The Sensory Profile has 125 items. Parents use a Likert scale to rate how frequently their child demonstrates a particular behavior (ranging from 1 = always to 5 = never). Total scale from 125-625, with a lower score indicates greater deviation from typically developing children and indicates more sensory reactivity symptoms.
Sensory Assessment for Neurodevelopmental Disorders (SAND) | After 12 weeks of growth hormone therapy
  A clinician-administered assessment and corresponding caregiver interview that is not dependent on verbal or cognitive ability and is therefore appropriate for severely affected or nonverbal individuals with PMS. Responses are rated by a trained examiner on an algorithm. Scores are dichotomous, 0 (not present) or 1 (present) and are based on a summary of observed sensory behaviors throughout the duration of the observation. A total SAND score ranging from 0 to 90. Higher scores represent a higher level of sensory reactivity symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kolevzon, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Seaver Autism Center for Research & Treatment, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data. Any purpose. Proposals should be directed to PI. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (tbd).

DOCUMENTS (1):
  • Informed Consent Form (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/77/NCT05187377/ICF_000.pdf